CLINICAL TRIAL: NCT03634072
Title: Pediatric REPlAcement of the PulmonaRy ValvE in Tetralogy of Fallot - The PREPARE-TOF Study
Brief Title: Pediatric REPlAcement of the PulmonaRy ValvE in Tetralogy of Fallot -
Acronym: TOFandPVR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to meet enrollment goal
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-015046; R34HL142142-01 (NIH)
Record Dates: First submitted 2018-08-02; First posted 2018-08-16 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Tetralogy of Fallot
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to PVR or no PVR
Who Masked: Investigator
Masking Description: Subjects will be randomly assigned to one of two groups. One will undergo PVR with catheter or surgery (whichever is most appropriate ). The other group will continue with medical management.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVR Arm (Other): PVR arm will undergo PVR via catheter or surgery
  Interventions: Procedure: PVR
- No PVR (No Intervention): No PVR group will continue with medical management

INTERVENTIONS:
Procedure: PVR — Subjects will undergo PVR via surgery or cardiac catheterization. PVR using cardiac catheterization may require a much shorter hospital stay than traditional heart surgery. If the valve is repaired by surgery, this will require open heart surgery to directly implant a pulmonary valve
  Arms: PVR Arm

SUMMARY:
Tetralogy of Fallot (TOF) is the most common cyanotic congenital heart defect with the vast majority of survivors of corrective surgery left with some degree of right ventricular (RV) volume overload due to pulmonary regurgitation (PR) which cause RV enlargement with right heart failure, diminished biventricular function, ventricular arrhythmia, sudden death and decreased exercise performance over time. Pulmonary valve replacement (PVR) has been thought to ameliorate these complications but the timing of replacement has yet to be determined with equipoise at the moment in this decision making process. As nearly all studies in this regard are retrospective with much less data in pediatric TOF than adults, this pilot trial sets the stage to create a prospective randomized trial in the teenage years.

DETAILED DESCRIPTION:
The purpose of this research study is to gather information on adolescents and young adults to help understand and improve the lives of patients with TOF.

Some patients diagnosed with TOF will have a procedure called pulmonary valve replacement (PVR) and some will not. PVR is done for valves that are too damaged to be repaired. This requires a surgeon or an expert in a procedure called cardiac catheterization to replace the damaged pulmonary valve with a valve made of tissue or a mechanical valve. Multiple studies in adult TOF patients have suggested that PVR may lessen many clinical symptoms but no one is sure if it truly does. There is little information about PVR in adolescence but it is thought that lessening the amount of leakage of the pulmonary valve at a young age may avoid future complications such as right heart failure or abnormal beats of your heart. There is no agreement among cardiologists, surgeons or other healthcare providers as to whether PVR truly helps avoid complications in the future and if it does, when PVR should be done. Using the information in this study, we hope to find out if PVR in adolescents is helpful in both the short and long term.

The Investigators believe the results of this study will help provide doctors with enough information to support a future large scale research study to further evaluate the outcomes PVR. This study will involve randomization to either the PVR or no PVR cohort, medical records review, exercise test and Cardiac Magnetic Resonance (CMR) , and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females with repaired Tetralogy of Fallot (TOF), currently between 13 and 21 years of age.
2. On clinical Cardiac Magnetic Resonance (CMR) : Right Ventricular End-Diastolic Volume Index (RVEDVi) between 140 and 180 cc/m2 inclusive with Right Ventricular End-Diastolic Function (RVEF) > 40% and Left Right Ventricular End-Diastolic (LVEF ) > 50%, RV outflow tract peak velocity < 3 meters/second (if not available this will be skipped); there will be no indexed Right Ventricular end-systolic volume (RVESVi) criteria; by defining RVEDVi and RVEF, Investigators will be inherently defining RVESVi
3. On clinical echocardiogram: RV outflow tract peak velocity < 3 meters/second (if not available this will be skipped), at least mild pulmonary insufficiency and tricuspid regurgitation with an RV pressure estimate < 1/2 systemic pressure.
4. On Exercise Stress Test (EST), aerobic capacity > 60% of predicted.
5. No Q-wave, R-wave, S-wave (QRS) duration criteria on ECG.

Exclusion Criteria:

1. Any condition judged by the patient's physician that would cause this trial to be detrimental to the patient.
2. Specific forms of TOF excluded are those with endocardial cushion defects, TOF with absent pulmonary valve and TOF with multiple aorto-pulmonary collaterals requiring unifocalization.
3. Unilateral branch pulmonary artery stenosis (one lung receives < 25% of total flow)
4. Contraindication to non-sedated exercise CMR (e.g. pacemaker/implanted cardioverter defibrillator); need for sedation
5. If data available, moderate or greater tricuspid regurgitation on echocardiogram or CMR or Qp/Qs > 1.5
6. Significant strokes/hemiplegia or inability to exercise
7. Genetic syndrome/developmental delay which would make QOL and EST date uninterpretable
8. Pregnancy
9. Previous pulmonary valve replacement (PVR)

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fogel, MD, Principal Investigator — The Childrens Hospital of Philadelphia
Locations (6):
- United States (6):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Cincinnati Children's Hosptial Medical Center, Cincinnati, Ohio
  - The Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The Principal Investigator (PI) is responsible for data management and accuracy of records. The PI may assign designated qualified individuals to collect the information. Only investigators' on this protocol and assigned research staff on this protocol will have access to the data. Data will be entered into a REDcap database by a member of the study team. All data and records generated during this study will be kept confidential in accordance with Institutional and HIPAA policies on subject privacy. The study team will not use such data and records for any purpose other than conducting the study. In order to keep protected health information from disclosure, each patient will be given a unique identification number. The key to this code will be kept in a locked file in one of the study investigator's offices. Any data that is transmitted to any Data Coordinating Center (DCC) will be de-identified by the enrolling site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2-3 years
Access Criteria: All future studies using these patients will require separate Institutional Review Board (IRB) approved protocols and consent forms. Only investigators' on this protocol and assigned research staff on this protocol will have access to the data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient was enrolled in 2020 in clinic
Pre-assignment Details: No pre-assignment issues were found
Groups:
- PVR Arm: PVR arm will undergo PVR via catheter or surgery
  PVR: Subjects will undergo PVR via surgery or cardiac catheterization. PVR using cardiac catheterization may require a much shorter hospital stay than traditional heart surgery. If the valve is repaired by surgery, this will require open heart surgery to directly implant a pulmonary valve.
  1 patient was enrolled in this arm from Emory University
- No PVR: No PVR group will continue with medical management
  No patients were enrolled in this group.
Period: Overall Study
Arm/Group | PVR Arm | No PVR
Started | 1 | 0
Completed | 0 (Study was terminated before completion) | 0
Not Completed | 1 | 0
Not completed — Early termination of overall study | 1 | 0

BASELINE CHARACTERISTICS:
Population: No patients enrolled in the No PVR group
Groups:
- Total: Total of all reporting groups
Arm/Group | PVR Arm | No PVR | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 17 (0) |  | 16 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Randomized to PVR Via Catheter or Surgery
Description: Participants will be randomized by computer by the statistician at the Data Coordinating Center (DCC) at Northwestern University (NU) who will maintain the schedule; this will be a 2:1 randomization of PVR to no-PVR. There will be no blinding and the assignment will not be concealed from the investigators. There will be no stratifications within each group.
Time Frame: 2-3 years
Population: One subject was randomized to the PVR arm; however, no data was collected to analyze
Measure: Number; unit: PVR via catheter or surgery
Arm/Group | PVR Arm | No PVR
Number analyzed (Participants) | 1 | 0
PVR via catheter or surgery | 0 |

2. Secondary Outcome: Exercise Performances
Description: This will be determined by exercise test performed to assess parameters such as oxygen consumption (VO2) at ventilatory anaerobic threshold (VAT) and normalized for age
Time Frame: 12-18 months
Population: No data were collected and no intervention completed in the PVR arm.
Arm/Group | PVR Arm | No PVR
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Prevalence of Arrhythmias
Description: This will be determined by reviewing Holter monitoring data to assess the prevalence of arrhythmias. This will also provide the endpoints for the larger, longer term trial
Time Frame: 12-18 months
Population: No data were collected and no intervention completed in the PVR arm.
Arm/Group | PVR Arm | No PVR
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Effects of Pulmonary Valve Replacement (PVR) on Diffuse Fibrosis
Description: This will be measured by obtaining preliminary data on the difference between patients randomized to PVR and no PVR in regard to diffuse fibrosis (DF).
Time Frame: 12-18 months
Population: No data were collected and no intervention completed in the PVR arm.
Arm/Group | PVR Arm | No PVR
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Effects of PVR on Exercise in the Magnetic Resonance (MR) Scanner
Description: Mechanisms of the effects of PVR in the definitive trial will be measured by obtaining preliminary data on the difference between patients randomized to PVR and no PVR in regard to performing exercise cardiac magnetic resonance (CMR).
Time Frame: 12-18 months
Population: No data were collected and no intervention completed in the PVR arm.
Arm/Group | PVR Arm | No PVR
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Effects of PVR on Biventricular Strain
Description: Mechanisms of the effects of PVR in the definitive trial will be measured by obtaining preliminary data on biventricular strain.
Time Frame: 12-18 months
Population: No data were collected and no intervention completed in the PVR arm.
Arm/Group | PVR Arm | No PVR
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Quality of Life (QOL)
Description: Quality of life will be measured using the Pediatric Cardiac Quality of Life Inventory (PCQLI) - to measure quality of life. The PCQLI has been used for over 10 years and is a validated quality of life metric. The PCQLI measures disease-specific, pediatric health related quality of life and generates 3 scores, namely, total, disease impact subscale, and psychosocial impact subscale. Each subscale score has a maximum of 50 points, and their sum yields the total score. Higher scores represent better perceived pediatric health related quality of life
Time Frame: 12-18 months
Population: No data were collected and no intervention completed in the PVR arm.
Arm/Group | PVR Arm | No PVR
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Only one patient enrolled in PVR arm. No adverse events (AEs) occurred.
Arm/Group | PVR Arm | No PVR
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Study terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03634072/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT03634072/ICF_001.pdf